CLINICAL TRIAL: NCT01564238
Title: Effect of Sodium Intake on Calcium Retention in Black and White Adolescent Girls.
Brief Title: Effect of Sodium Intake on Calcium Retention in Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Institute of Child Health (Other)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Camp Calcium 5-6
Record Dates: First submitted 2012-02-02; First posted 2012-03-27 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: calcium retention; sodium retention
MeSH Terms: conditions — Osteoporosis; Hypernatremia | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High calcium diets (1300 mg or higher) (Experimental)
  Interventions: Other: Low Na diet (1.3 g/d); Other: High sodium diet (3.8 g/d)
- Low calcium diet (800 mg/d) (Experimental)
  Interventions: Other: Low Na diet (1.3 g/d); Other: High sodium diet (3.8 g/d)

INTERVENTIONS:
Other: Low Na diet (1.3 g/d) — 20 day controlled feeding study (live in) providing 1.3 grams per day of sodium.
  Other Names: low sodium; sodium calcium
Other: High sodium diet (3.8 g/d) — 20 day controlled feeding study (live in) providing 3.8 grams per day of sodium.
  Other Names: high sodium; sodium calcium

SUMMARY:
Optimal calcium retention is important for building bone mass within the genetic potential, a key to reducing risk of osteoporosis later in life. Calcium retention is high during the rapid growth period. The investigators know that urinary calcium is affected by sodium intake but the investigators do not know the effects of sodium intake during the growth spurt or the differences in calcium retention between blacks and whites. Our hypothesis was that a high dietary sodium increases the calcium intakes required for optimal calcium retention in both black and white adolescent girls. The investigators tested calcium retention while girls consumed a low and high sodium diet during three week periods. The subjects were housed in a Purdue fraternity house during the summer and they were supervised at all times by trained staff. During the summer of 1999, subjects consumed diets with 2 levels of dietary Na+ with a fixed diet low in calcium. On the next summer, they switched to a high calcium diet. Subjects collected fecal and urine daily for 20 days. Other measurements included daily body weight, blood pressure every other day, blood sample at the end of each session. Baseline measures included bone mass, self-assessment of pubertal development, a physical examination and diet history.

DETAILED DESCRIPTION:
Optimal calcium retention is a prerequisite for building maximal peak bone mass within the genetic potential, a key to reducing risk of osteoporosis later in life. The investigators have determined that maximal calcium retention averages 423 mg/day during the period of rapid skeletal accretion in white girls at a mean dietary calcium intake of 1300 mg/d. Urinary calcium explains more than 50% of the variance in calcium retention. However, urinary sodium (i.e. sodium intake)is a major determinant of urinary calcium excretion and the effect of sodium intake on maximal calcium retention is not known. Nor is its effect known in black adolescents who have higher bone density and lower calcium excretion than white adolescents.

The primary aim was to test the hypothesis that high dietary sodium increases the calcium intakes required for optimal calcium retention in both black and white adolescent girls. Calcium retention was measured at two levels of dietary sodium in a randomized crossover design on one of two levels of dietary calcium intake in black and white adolescent girls during three week metabolic periods. The investigators hypothesized that the mechanisms which regulate sodium reabsorption in the renal tubules also regulate calcium retention. Increased incidence of hypertension in blacks compared to whites has been attributed to increased sodium retention. Sodium intake induced changes in calcium and sodium retention in both races were related to changes in sodium handling (plasma renin activity, serum aldosterone, and salt sensitivity) and calcium regulating hormones, biomarkers of bone turnover and bone mass.

The subjects were resident in a Purdue fraternity house, which was transformed during the summer into a metabolic unit. Subjects were supervised at all times by trained staff. The balance study was divided into 2 sessions of 3 weeks each during the summer of 1999 and 2000, with 2 levels of dietary Na+ during each summer. During the summer of 1999 subjects consumed a low calcium diet while in the summer of 2000 subjects consumed a high calcium diet. The Na+ intake periods were separated by a 2-week period, in which subjects were free to consume self-selected diets. Subjects collected fecal and urine daily for 20 days. Other measurements included daily body weight, blood pressure every other day, blood sample at the end of each session. Baseline measures included bone mass, self-assessment of pubertal development, a physical examination and diet history.

ELIGIBILITY:
Inclusion Criteria:

* White or black race (both parents and grandparents had to be white or black to be eligible in the study).

Exclusion Criteria:

* < 11 or > 15 years
* body mass index (BMI) of < 15th or > 85th percentile for age
* history of amenorrhea, pregnancy or abortion, eating disorders, oral contraceptive or tobacco use.

Ages: 11 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 1999-01; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Change in calcium retention(mg/d)due to high (4g/d) and low (1g/d) sodium intake. | Up to 12 weeks

SECONDARY OUTCOMES:
Potassium retention in the black and white adolescent subjects | Up to 12 weeks
Racial differences on the effects of high and low sodium intake levels on calcium intake requirements and calcium retention in adolescent girls | Up to 12 weeks
Magnesium retention in the black and white adolescent subjects | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Purdue University; Berdine R Martin, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Result] Palacios C, Wigertz K, Martin BR, Braun M, Pratt JH, Peacock M, Weaver CM. Racial differences in potassium homeostasis in response to differences in dietary sodium in girls. Am J Clin Nutr. 2010 Mar;91(3):597-603. doi: 10.3945/ajcn.2009.28400. Epub 2009 Dec 9. PMID 20007307
- [Result] Thierry-Palmer M, Henderson VM, Hammali RE, Cephas S, Palacios C, Martin BR, Weaver CM. Black and white female adolescents lose vitamin D metabolites into urine. Am J Med Sci. 2008 Apr;335(4):278-83. doi: 10.1097/MAJ.0b013e31815768db. PMID 18414066
- [Result] Braun M, Palacios C, Wigertz K, Jackman LA, Bryant RJ, McCabe LD, Martin BR, McCabe GP, Peacock M, Weaver CM. Racial differences in skeletal calcium retention in adolescent girls with varied controlled calcium intakes. Am J Clin Nutr. 2007 Jun;85(6):1657-63. doi: 10.1093/ajcn/85.6.1657. PMID 17556706
- [Result] Wigertz K, Palacios C, Jackman LA, Martin BR, McCabe LD, McCabe GP, Peacock M, Pratt JH, Weaver CM. Racial differences in calcium retention in response to dietary salt in adolescent girls. Am J Clin Nutr. 2005 Apr;81(4):845-50. doi: 10.1093/ajcn/81.4.845. PMID 15817862
- [Result] Palacios C, Wigertz K, Martin BR, Jackman L, Pratt JH, Peacock M, McCabe G, Weaver CM. Sodium retention in black and white female adolescents in response to salt intake. J Clin Endocrinol Metab. 2004 Apr;89(4):1858-63. doi: 10.1210/jc.2003-031446. PMID 15070956
- [Derived] Palacios C, Wigertz K, Braun M, Martin BR, McCabe GP, McCabe L, Pratt JH, Peacock M, Weaver CM. Magnesium retention from metabolic-balance studies in female adolescents: impact of race, dietary salt, and calcium. Am J Clin Nutr. 2013 May;97(5):1014-9. doi: 10.3945/ajcn.112.039867. Epub 2013 Apr 3. PMID 23553157